CLINICAL TRIAL: NCT01080144
Title: A Pilot Study Aiming to Assess the Feasibility of Critical Flicker Frequency for the Diagnosis of Minimal Encephalopathy in Patients With Cirrhosis
Brief Title: Feasibility of Critical Flicker Frequency Procedure for the Diagnosis of Minimal Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09 156 02
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; TIPS (Transjugular intrahepatic portosystemic shunt); Encephalopathy
MeSH Terms: conditions — Fibrosis; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Critical Flicker Frequency (Experimental): Critical Flicker Frequency Procedure
  Interventions: Other: Critical flicker frequency procedure

INTERVENTIONS:
Other: Critical flicker frequency procedure — After TIPS, patients will be followed during one year and the psychometric test and Critical flicker frequency procedure will be performed every 3 months

SUMMARY:
All patients eligible for TIPS (Transjugular intrahepatic portosystemic shunt) procedure will be considered for inclusion. After written inform consent, psychometric tests in order to calculate the psychometric hepatic encephalopathy (PHES) score, the gold standard for the diagnosis of minimal encephalopathy and critical flicker frequency (CFF) will be performed before the TIPS procedure. After TIPS, patients will be followed during one year and the psychometric test and CFF will be performed every 3 months.

30 patients will be included.

The main endpoint is the success rate of CFF. The secondary end points are

* Correlation between CFF and PHES score
* Performance of CFF and PHES score to predict the occurrence of overt encephalopathy after TIPS procedure
* A sample collection during TIPS procedure is also performed for validation of biomarkers

ELIGIBILITY:
Inclusion Criteria:

* patients with cirrhosis in whom a TIPS is indicated
* patients have given their informed consent te be included

Exclusion Criteria:

* minor
* pregnant women
* patients who cannot see the red color
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
success rate of Critical Flicker Frequency (CFF) Procedure | before TIPS and every 3 months till one year
  number of patients in whom ten measurement will be available / 30 patients

SECONDARY OUTCOMES:
occurrence of encephalopathy | every 3 months till one year after TIPS procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Bureau, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Dr Christophe Bureau, Toulouse, Hôpital Rangueil, France

REFERENCES:
- [Result] Berlioux P, Robic MA, Poirson H, Metivier S, Otal P, Barret C, Lopez F, Peron JM, Vinel JP, Bureau C. Pre-transjugular intrahepatic portosystemic shunts (TIPS) prediction of post-TIPS overt hepatic encephalopathy: the critical flicker frequency is more accurate than psychometric tests. Hepatology. 2014 Feb;59(2):622-9. doi: 10.1002/hep.26684. PMID 24620380